CLINICAL TRIAL: NCT02742454
Title: VentFirst: A Multicenter RCT of Assisted Ventilation During Delayed Cord Clamping for Extremely Preterm Infants
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Virginia (Other)
Collaborators: Brigham and Women's Hospital (Other); Mayo Clinic (Other); St. Louis University (Other); University of Colorado, Denver (Other); Oregon Health and Science University (Other); University of Calgary (Other); Columbia University (Other); Indiana University (Other); University of California, Davis (Other); University of Alberta (Other); University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Karen Fairchild, MD, Professor of Pediatrics, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 18783
Record Dates: First submitted 2016-04-14; First posted 2016-04-19 (Estimated); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: Intraventricular Hemorrhage
Keywords: Umbilical Cord Clamping; Intraventricular Hemorrhage; Extremely Preterm Infants

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Board-certified radiologists interpreting head ultrasound findings are blinded to study arm. Consensus on maximum grade of IVH between two radiologists (some combination of site radiologist and one of three external readers blinded to each others' interpretation) is required.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard 30-60 Seconds Cord Clamping (Active Comparator): Standard treatment for extremely preterm infants which is delayed cord clamping 30-60 seconds after birth, and assisted ventilation after cord clamping.
  Interventions: Procedure: Standard 30-60 Seconds Cord Clamping
- VentFirst 120 Seconds Cord Clamping (Experimental): Assisted ventilation (face mask continuous positive airway pressure, CPAP, or positive pressure ventilation, PPV) is provided prior to cord clamping at 120 seconds.
  Interventions: Procedure: VentFirst 120 Seconds Cord Clamping

INTERVENTIONS:
Procedure: Standard 30-60 Seconds Cord Clamping — The infant is stimulated to breathe after birth. If the infant is not breathing well, the cord is clamped at 30 seconds. If the baby is breathing well, the cord is clamped at 60 seconds. Ventilatory assistance is given after cord clamping.
  Arms: Standard 30-60 Seconds Cord Clamping
Procedure: VentFirst 120 Seconds Cord Clamping — The infant is stimulated to breathe after birth. If the infant is not breathing well, PPV by face mask is given starting at 30 seconds. If the baby is breathing well, CPAP is given starting at 30 seconds. The cord is clamped at 120 seconds.
  Arms: VentFirst 120 Seconds Cord Clamping

SUMMARY:
The purpose of this study is to determine whether providing ventilatory assistance prior to umbilical cord clamping influences the occurrence of intraventricular hemorrhage (IVH) in extremely preterm (EPT) infants, compared to standard care of providing ventilatory assistance after cord clamping.

DETAILED DESCRIPTION:
Newborns with gestational age 23 wks 0 days through 28 wks 6 days are randomized to control (delayed cord clamping for at least 30 seconds, or up to 60 seconds if breathing spontaneously, with ventilatory assistance provided after) or the VentFirst intervention (ventilatory assistance with continuous positive airway pressure or positive pressure ventilation given starting 30 seconds after birth and cord clamping at 120 seconds).

The primary outcome is lack of IVH on 7-10 day head ultrasound or death before day 7.

The study was designed to test the impact of the intervention in each of two cohorts:

1. Infants not breathing well 30 seconds after birth
2. Infants breathing well 30 seconds after birth

Randomization and analysis is stratified by gestational age category:

1. 23 0/6 to 25 6/7 weeks' gestation
2. 26 0/7 to 28 6/7 weeks' gestation

ELIGIBILITY:
Inclusion Criteria:

* 23 0/7 - 28 6/7 weeks' gestation at delivery

Exclusion Criteria:

* Life-threatening condition of fetus (e.g. severe hydrops, lethal chromosomal abnormality, severe congenital malformation)
* Suspected severe fetal anemia
* Monochorionic or monoamniotic twins
* Multiple gestation greater than twins
* Decision made for comfort care only
* Medical emergency necessitating emergency delivery (e.g. complete placental abruption)
* Obstetrician or Neonatology concern for inappropriateness of the study intervention based on maternal or fetal factors.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 570 (Actual)
Dates: Start 2016-06; Primary Completion 2023-03 (Actual); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Intraventricular Hemorrhage on Head Ultrasound or death before 7 days of age | 7-10 days after birth
  presence of any grade IVH on HUS

SECONDARY OUTCOMES:
5 minute Apgar Score <5 | 5 minutes after birth
  Low Apgar score (<5) at 5 minutes
Lowest hematocrit in first 24 hours | First 24 hours after birth
  Median, 25th & 75th percentiles
Medication for low blood pressure in first 24 hours | First 24 hours after birth
  Hydrocortisone and/or vasopressor for hypotension
Number of red blood cell transfusions birth through day 10 | First 10 days after birth
  Median, 25th & 75th percentiles
Severe brain injury on head ultrasound | Birth through 36 weeks' postmenstrual age
  Grade 3-4 IVH and/or cerebellar hemorrhage and/or cystic periventricular leukomalacia on head ultrasound at 7-10 days of age and/or near 36 weeks' postmenstrual age
Death | Birth through 36 weeks' postmenstrual age
  All-cause mortality

OTHER OUTCOMES:
Maternal post-partum hemorrhage | First 24 hours after delivery
  >= 1000 mL estimated blood loss
Maternal red blood cell transfusion | Prior to maternal hospital discharge
  Administration of an RBC transfusion
Maternal retained placenta | Prior to hospital discharge
  Retained placenta
Maternal post-partum delivery related infection | Prior to maternal hospital discharge
  Diagnosis of a delivery related infection
Apgar scores | 1 minute, 5 minutes, and 10 minutes after delivery
  Apgar scores taken in the delivery room (1, 5, 10 minutes)
Umbilical Cord Blood Gas | In delivery room
  Umbilical cord venous and arterial pH
Chest compressions or epinephrine | In delivery room
  occurrence of infant chest compressions or administration of epinephrine
Volume Bolus | In delivery room
  administration of a volume bolus
Intubation | In delivery room
  Endotracheal intubation
Admission hypothermia <36.5°C | at admission to the Neonatal Intensive Care Unit
  <36.5°C
Pneumothorax | first 24 hours after delivery
  Diagnosis of pneumothorax requiring intervention
NICU admission temperature | At NICU admission
  Infant's NICU admission temperature
SNAPPE-II Score | First 12 hours after birth
  Score for Neonatal Acute Physiology-Perinatal Extension
Red blood cell transfusion | First 24 hours after birth
  Administration of an RBC transfusion
Highest hematocrit | First 24 hours after birth
  Infant's highest hematocrit (before transfusion)
Lowest mean arterial blood pressure | First 24 hours after birth
  Infant's lowest mean arterial blood pressure (cuff or arterial catheter)
Volume Bolus | First 24 hours after birth
  Any volume bolus including the delivery room, and including NICU packed red blood cells, platelets, plasma, saline, or other fluid bolus
Surfactant administration | First 10 days after birth
  Administration of surfactant
Mechanical ventilation days | First 10 days after birth
  Number of days on mechanical ventilation via an endotracheal tube
Early-Onset Septicemia | <72 hours after birth
  Positive blood culture in first 3 days and treated with at least 5 days of antibiotics
Highest bilirubin | First 10 days after birth
  Highest bilirubin recorded
Phototherapy duration | First 10 days after birth
  Number of days on phototherapy
Intraventricular hemorrhage | Prior to 36 weeks' postmenstrual age
  Highest grade of IVH
Cerebellar hemorrhage | Prior to 36 weeks' postmenstrual age
  occurrence of cerebellar hemorrhage
Late-Onset Septicemia | Prior to 36 weeks' postmenstrual age
  Positive blood culture after first 3 days and treated with at least 5 days of antibiotics
Cystic Periventricular Leukomalacia (cPVL) | Prior to 36 weeks' postmenstrual age
  Occurrence of cPVL
Patent Ductus Arteriosus (PDA) | Prior to 36 weeks' postmenstrual age
  occurrence of PDA requiring pharmacological or surgical treatment
Spontaneous intestinal perforation (SIP) | Prior to 36 weeks' postmenstrual age
  SIP without NEC and requiring surgery or peritoneal drain
Necrotizing Enterocolitis (NEC) | Prior to 36 weeks' postmenstrual age
  Occurrence of NEC modified Bell's stage 2-3
Bronchopulmonary Dysplasia (BPD) | At 36 weeks' postmenstrual age
  Occurrence of BPD receiving continuous supplemental oxygen
Severe ROP | Prior to 36 weeks' postmenstrual age
  occurrence of ROP stage 3 or treated with laser or bevacizumab

CONTACTS AND LOCATIONS:
Overall Officials: Karen Fairchild, MD, Principal Investigator — University of Virginia
Locations (12):
- United States (10):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of California, Davis, Sacramento, California
  - University of Colorado, Denver, Colorado
  - University of Indiana, Indianapolis, Indiana
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - St. Louis University, St Louis, Missouri
  - Columbia University Medical Center, New York, New York
  - Oregon Health & Science University, Portland, Oregon
  - University of Virginia, Charlottesville, Virginia
- Canada (2):
  - University of Calgary, Calgary, Alberta
  - University of Alberta, Edmonton, Edmonton, Alberta

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fang JL, Fairchild KD, Petroni GR, Strand ML, Warren JB, Law BH, Gorman TE, Leone TA, Thomas SP, Niermeyer S; VentFirst Consortium. Physiologic Transition During Delayed Cord Clamping With Assisted Ventilation in Preterm Infants: A Secondary Analysis of the VentFirst Trial. JAMA Netw Open. 2025 Nov 3;8(11):e2545258. doi: 10.1001/jamanetworkopen.2025.45258. PMID 41284295
- [Derived] Fairchild KD, Petroni GR, Varhegyi NE, Strand ML, Josephsen JB, Niermeyer S, Barry JS, Warren JB, Rincon M, Fang JL, Thomas SP, Travers CP, Kane AF, Carlo WA, Byrne BJ, Underwood MA, Poulain FR, Law BH, Gorman TE, Leone TA, Bulas DI, Epelman M, Kline-Fath BM, Chisholm CA, Kattwinkel J; VentFirst Consortium. Ventilatory Assistance Before Umbilical Cord Clamping in Extremely Preterm Infants: A Randomized Clinical Trial. JAMA Netw Open. 2024 May 1;7(5):e2411140. doi: 10.1001/jamanetworkopen.2024.11140. PMID 38758557